CLINICAL TRIAL: NCT03916146
Title: Behavioral Parent Training for Families With Deaf and Hard of Hearing Preschoolers
Acronym: CHAMPS-DHH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christina Studts (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor-Investigator, Christina Studts, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 45213; R01DC016957 (NIH)
Record Dates: First submitted 2019-04-11; First posted 2019-04-16 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Deafness; Hearing Loss; Parenting; Child Behavior
MeSH Terms: conditions — Deafness; Hearing Loss; Child Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral Parent Training (Experimental)
  Interventions: Behavioral: Parent Training Intervention
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Parent Training Intervention — Adapted version of the Family Check-Up/Everyday Parenting intervention
  Arms: Behavioral Parent Training

SUMMARY:
Children who are deaf and hard of hearing (DHH) rarely receive behavioral interventions to prevent the long-term costly outcomes of behavior problems. This project will systematically adapt an evidence-based parent training intervention to increase its acceptability and relevance for parents of young DHH children. Effectiveness of the adapted intervention and its implementation with parents of young DHH children followed in "real world" hearing healthcare clinics will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Parent is age 18 or older
* Parent is custodial guardian of child
* Parent can either speak/understand English or use American Sign Language
* Parent lives in a state with an established referral network for parents of DHH children if additional services are needed
* At baseline, child is between the ages of 3 and 6 years
* At baseline, child lives majority of time in the parent/guardian's home
* Child is deaf or hard of hearing
* Child has used hearing aid(s), cochlear implant(s) and/or bone conduction device(s) for greater than 6 months

Exclusion Criteria:

* Active child protective services case is open
* Parent has already accessed behavioral health services for the child
* Parent participated in formative research for this study

Ages: 3 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2020-01-31 (Actual); Primary Completion 2024-10-14 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Parenting Young Children (PARYC) Scale | 6 months after parent baseline
  parent self-report of use of positive parenting strategies

SECONDARY OUTCOMES:
Child Behavior Checklist (CBCL) | 6 months, 12 months, 18 months, 24 months, 30 months, 36 months after parent baseline
  subscale and total scores
Parent Sense of Competence Scale (PSCS) | 6 months, 12 months, 18 months, 24 months, 30 months, 36 months after parent baseline
  parent-report self-efficacy and satisfaction with the parenting role
Parent Child Interaction System (PARCHISY) | 12 months, 24 months, 36 months after parent baseline
  observational measure of parent-child interaction quality
Beck Depression Inventory-II (BDI-II) | 6 months, 12 months, 18 months, 24 months, 30 months, 36 months after parent baseline
  parent-report depressive symptoms
Parent Motivation Inventory (PMI) | 12 months, 24 months, 36 months after parent baseline
  parent-report motivation to change parenting behaviors
Therapy Attitude Inventory (TAI) | 6 months, 18 months, 30 months after parent baseline
  parent-report satisfaction with intervention
Hearing Aid Adherence Questionnaire | 12 months, 24 months, 36 months after parent baseline
  parent-report use of hearing aids by child
Change in Parenting Young Children scale (PARYC) scores over time | 6 months, 12 months, 18 months, 24 months, 30 months, 36 months after parent baseline
  While the primary study outcomes is PARYC scores 6 months after baseline, we will also assess differences in changes over 3 years in PARYC scores within and between study arms

OTHER OUTCOMES:
Data-logging of hearing aid/cochlear implant use by child | 12 months, 24 months, 36 months after parent baseline
  as available from audiological medical records
MacArthur Bates Communicative Development Inventories | 12 months, 24 months, 36 months after parent baseline
  parent-report of children's developing abilities in early language
Peabody Picture Vocabulary Test (PPVT) | 12 months, 24 months, 36 months after parent baseline
  measure of child's receptive language
Clinical Evaluation of Language Fundamentals - Preschool | 12 months, 24 months, 36 months after parent baseline
  assessment of language pragmatics for children
Beginner's Intelligibility Test (BIT) | 12 months, 24 months, 36 months (children ages 3 years +) after parent baseline
  assessment of child's intelligibility
Meaningful Auditory Integration Scale (MAIS) | 12 months, 24 months, 36 months after parent baseline
  parent report of child's language skills in real-world situations

CONTACTS AND LOCATIONS:
Overall Officials: Christina Studts, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made publicly available (by request to the PI) immediately following the acceptance for publication of the main findings from the final dataset.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: De-identified data will be made publicly available (by request to the PI) immediately following the acceptance for publication of the main findings from the final dataset.
Access Criteria: De-identified data will be made publicly available (by request to the PI) immediately following the acceptance for publication of the main findings from the final dataset.

DOCUMENTS (1):
  • Informed Consent Form (2023-02-01): https://cdn.clinicaltrials.gov/large-docs/46/NCT03916146/ICF_000.pdf